CLINICAL TRIAL: NCT00005067
Title: A Phase I Trial of Photodynamic Therapy With Lutetium Texaphyrin in Patients With Locally Recurrent Prostate Carcinoma
Brief Title: Photodynamic Therapy With Lutetium Texaphyrin in Treating Patients With Locally Recurrent Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02323; UPCC 6899; CDR0000067672 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — motexafin lutetium; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

ARMS (1):
- Treatment (motexafin lutetium, PDT) (Experimental): Patients receive lutetium texaphyrin IV over 10-15 minutes 3-24 hours before photodynamic therapy (PDT). Optical fibers attached to a laser are inserted through a catheter into the prostate. The laser delivers 730 nm light to the prostate until the specified fluence is delivered. Patients undergo biopsy of the prostate and bladder before and after PDT. Cohorts of 3-6 patients receive escalating doses of lutetium texaphyrin and light fluence until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.
  Interventions: Drug: motexafin lutetium; Drug: photodynamic therapy

INTERVENTIONS:
Drug: motexafin lutetium — Given IV
  Other Names: Antrin; lutetium texaphrin; lutetium texaphyrin; Lutex; PCI-0123
Drug: photodynamic therapy — Undergo photodynamic therapy
  Other Names: Light Infusion Therapy™; PDT; therapy, photodynamic

SUMMARY:
This phase I trial is studying the side effects and best dose of photodynamic therapy with lutetium texaphyrin in treating patients with locally recurrent prostate cancer. Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. This may be effective treatment for locally recurrent prostate cancer. Photosensitizing drugs, such as lutetium texaphyrin, are absorbed by cancer cells and, when exposed to light, become active and kill the cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose limiting toxicities and maximum tolerated dose of photodynamic therapy (PDT) using 730 nm light and lutetium texaphyrin in patients with locally recurrent prostate adenocarcinoma who have failed previous definitive radiotherapy.

SECONDARY OBJECTIVES:

I. Measure lutetium texaphyrin levels in needle biopsies of the prostate before and after PDT using an HPLC and tissue fluorescence assay and calculate the percent change in lutetium texaphyrin after treatment.

II. Measure lutetium texaphyrin fluorescence in situ in the prostate before and after PDT using optical methods and correlate these results with the direct tissue measurements made in the biopsies of these patients.

III. Determine clinical outcome including clinical response, progression free survival, time to complete response, time to biochemical relapse, time to local progression, time to distant failure, overall survival, and disease specific survival in these patients treated with this regimen.

OUTLINE: This is a dose-escalation study of lutetium texaphyrin and light fluence.

Patients receive lutetium texaphyrin IV over 10-15 minutes 3-24 hours before photodynamic therapy (PDT). Optical fibers attached to a laser are inserted through a catheter into the prostate. The laser delivers 730 nm light to the prostate until the specified fluence is delivered. Patients undergo biopsy of the prostate and bladder before and after PDT. Cohorts of 3-6 patients receive escalating doses of lutetium texaphyrin and light fluence until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

Patients are followed at 2 weeks, 1 month, 2 months, 3 months, then every 3 months until 2 years, then every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 24 patients will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally recurrent prostate adenocarcinoma previously treated with definitive radiotherapy
* No T3 or T4 primary tumors
* No evidence of regional or distant metastases by MRI or bone scan
* No pathologic demonstration of malignancy in pelvic or abdominal lymph nodes
* Prostate gland volume no greater than 50 mL by MRI or ultrasound
* PSA no greater than 20 ng/mL
* Performance status - ECOG 0-2
* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* No severe liver disease (e.g., cirrhosis or grade III-IV elevations in liver function studies)
* Bilirubin no greater than 1.5 mg/dL
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* Medical suitability for implantation
* Fertile patients must use effective contraception during and for 6 months after study participation
* No history of grade III or IV genitourinary or gastrointestinal toxicity
* No known G6PD deficiency
* No porphyria
* At least 4 weeks since prior gene therapy
* At least 4 weeks since prior immunotherapy
* At least 4 weeks since prior combination chemotherapy
* No concurrent chemotherapy
* At least 4 weeks since prior hormonal therapy
* No concurrent hormonal therapy
* No prior cryosurgery for prostate cancer
* No other concurrent medication for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2000-02; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) defined as grade III non-hematologic toxicity or grade IV hematologic toxicity as assessed by the Cancer Therapy Evaluation Program Common Toxicity Criteria (CTC) version 2.0 | 24 hours
MTD based on the incidence of DLT as assessed by the Cancer Therapy Evaluation Program CTC version 2.0 | 24 hours

SECONDARY OUTCOMES:
Percent change in lutetium texaphyrin levels in needle biopsies by high pressure liquid chromatography (HPLC) and tissue fluorescence assay | From pre-PDT to post-PDT
  Scattergrams and error bar plots of lutetium texaphyrin concentration by lutetium texaphyrin dose level and possibly by light fluence (for a fixed lutetium texaphyrin dose = 2) will be constructed to investigate possible dose-concentration relationships.
Lutetium texaphyrin levels in situ | At pre- and post-PDT
  Descriptive statistics (mean, median, standard deviation, range and coefficient of variation) will be used to characterize the distribution of lutetium texaphyrin concentrations within each dose level.
Clinical response rate defined as no evidence of disease (NED) | Up to 5 years
  The 95% confidence interval will be calculated for the rate of NED.
Progression-free survival (PFS) | From the date of accession to the date of documentation of clinical progression or until the date of death from any cause, assessed up to 5 years
  Estimated by the method of Kaplan and Meier.
Time to complete response | Up to 5 years
Time to biochemical relapse | Up to 5 years
Time to local progression as determined by clinical exam | From the date of accession to the date of documented local progression, assessed up to 5 years
  Estimated by the method of Kaplan and Meier.
Time to distant failure | From the date of accession to the date of documented metastatic disease, assessed up to 5 years
Overall survival | From the date of accession to the date of death, assessed up to 5 years
Disease specific survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Michael Hahn, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States